CLINICAL TRIAL: NCT03783858
Title: Image Collection of Normal Eyes on the Optos P200TE for Development of an EU Reference Database
Brief Title: Image Collection of Normal Eyes for Development of an EU RDB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPT1030
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single (Other)
  Interventions: Device: P200TE

INTERVENTIONS:
Device: P200TE — OCT images

SUMMARY:
This study is designed to collect in-tissue OCT scans on the Optos P200TE on normal healthy eyes to develop a EU reference database

ELIGIBILITY:
Inclusion Criteria:

1. Subject 22 years of age or older on the date of informed consent
2. Subject able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subject presenting at the site with normal eyes* (Cataracts and LASIK and PRK are allowed)
4. BCVA 20/40 or better (each eye)
5. Subject is able to comply with the study procedures in the view of the investigator *Normal eyes are defined as eyes judged normal for the subjects age as determined by the PI or sub-investigator

Exclusion Criteria:

1.1. Subject unable to tolerate ophthalmic imaging 2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images 3. History of leukemia, dementia or multiple sclerosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Retinal thickness | 1 day
  In general, descriptive statistics (n, mean, standard deviation, median, minimum and maximum) and 95% confidence interval for the mean will be used to summarize each scan parameters.
  The 1st, 5th, 95th and 99th percentile results will be tabulated. All percentile results will be incorporated in the device software.

CONTACTS AND LOCATIONS:
Overall Officials: Tunde Peto, PhD, Principal Investigator — Queens University Belfast
Locations (5):
- United Kingdom (5):
  - Simon Browning Optometrist, Bedford, England
  - Barnard Levit Optometrists, London, England
  - London Vision Clinic, London, England
  - Queens University, Belfast, Northern Ireland
  - Cameron Optometry, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: No